CLINICAL TRIAL: NCT04817332
Title: A Randomised Double-blind Placebo-controlled Trial of Brensocatib (INS1007) in Patients With Severe COVID-19
Brief Title: STOP-COVID19: Superiority Trial Of Protease Inhibition in COVID-19
Acronym: STOP-COVID19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Dundee (Other)
Collaborators: NHS Tayside (Other Government); Insmed Incorporated (Industry)
Responsible Party: Principal Investigator, James Chalmers, Professor of Respiratory Research, University of Dundee
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01.01.20; 2020-001643-13 (EudraCT Number); 281986 (Other: IRAS)
Record Dates: First submitted 2021-01-25; First posted 2021-03-26 (Actual); Results first posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — brensocatib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Brensocatib (Experimental): Brensocatib oral tablet, 25mg once per day for 28 days
  Interventions: Drug: Brensocatib
- Placebo (Placebo Comparator): Placebo oral tablet, 25mg once per day for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brensocatib — Selective, competitive, and reversible inhibitor of DPP1
  Other Names: INS1007
  Arms: Brensocatib
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
COVID-19 is a respiratory disease caused by a novel coronavirus (SARS-CoV-2) and causes substantial morbidity and mortality. There is currently no vaccine to prevent infection with SARS-CoV-2 and no therapeutic agent to treat COVID-19. This clinical trial is designed to evaluate the potential of Brensocatib (INS1007) as a novel host directed therapy for the treatment of adult patients hospitalized with COVID-19. The investigators hypothesise that Brensocatib, by blocking damaging neutrophil proteases, will reduce the incidence of acute lung injury and acute respiratory distress syndrome (ARDS) in patients with COVID-19, thereby resulting in improved clinical outcomes at day 15 and day 29, fewer days dependent on oxygen or mechanical ventilation, and shorter length of hospital stay.

High rates of patients requiring mechanical ventilation and overwhelming intensive care unit capacity has been the major issue contributing to excess deaths in Italy and Spain during the pandemic and is likely to be a major issue in other countries such as the United Kingdom in the coming weeks. Treatments that could prevent the requirement for mechanical ventilation or shorten the duration of ICU stay by reducing the severity of ARDS are therefore the number 1 target for COVID19 therapy.

The investigators recently conducted a large phase 2 study of Brensocatib in patients with bronchiectasis designed to test if treatment with Brensocatib could reduce infective exacerbations and reduce neutrophil elastase activity in the lung in bronchiectasis patients. The study met its primary endpoint of time to first exacerbation and key secondary endpoint of the frequency of exacerbations as well as showing marked reductions in neutrophil elastase concentrations in sputum.

Participants will be randomised to receive Brensocatib or placebo 25mg orally once daily for 28 days.

DETAILED DESCRIPTION:
BACKGROUND COVID-19 is a respiratory disease caused by a novel coronavirus severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2) and causes substantial morbidity and mortality.This clinical trial is designed to evaluate the potential of Brensocatib as a novel host directed therapy for the treatment of adult patients hospitalised with COVID-19. The investigators hypothesise that Brensocatib, by blocking damaging neutrophil proteases, will reduce the incidence of acute lung injury and acute respiratory distress syndrome (ARDS) in patients with COVID-19, thereby resulting in improved clinical outcomes at day 15 and day 29, fewer days dependent on oxygen or mechanical ventilation, and shorter length of hospital stay.

Coronavirus (CoVs) are positive-sense single stranded enveloped Ribonucleic acid (RNA) viruses, many of which are commonly found in humans and cause mild symptoms. Over the past two decades, emerging pathogenic CoVs capable of causing life-threatening disease in humans and animals have been identified, namely severe acute respiratory syndrome (SARS) coronavirus (SARS-CoV) and Middle Eastern respiratory syndrome coronavirus (MERS- CoV).

In December 2019, the Wuhan Municipal Health Committee (Wuhan, China) identified an outbreak of viral pneumonia cases of unknown cause.5 Coronavirus RNA was quickly identified in some of these patients. This novel coronavirus has been abbreviated as SARS-COV-2 and has 89% nucleotide identity with bat SARS-like-CoVZXC21 and 82% with that of human SARS-CoV. This novel coronavirus has been designated SARS-CoV-2, and the disease caused by this virus has been designated COVID-19. Initial infections were travel associated with individuals having contact with Wuhan or other affected areas but the disease has now spread to affect hundreds of thousands of patients worldwide with widespread community transmission across the globe.

Outbreak forecasting and mathematical modelling suggest that these numbers will continue to rise.

Global efforts to evaluate novel antivirals and therapeutic strategies to treat COVID-19 have intensified but to date dexamethasone is the only therapy shown to reduce mortality in COVID-19 while repurposed antiviral drugs did not show clinical benefits in the World Health Organisation SOLIDARITY trial.

Mortality from COVID-19 has been estimated at between 0.5% and 3.4% of infected patients and occurs most frequently because of the development of ARDS. In contrast to some, particularly bacterial pneumonias, where patients present with acute respiratory failure and sepsis, the dynamics of COVID-19 infection demonstrate a slow deterioration in oxygenation with the development of bilateral infiltrates in a high proportion of patients, consistent with the development of ARDS. Patients subsequently require mechanical ventilation.

Treatments that could prevent the requirement for mechanical ventilation or shorten the duration of intensive care unit stay by reducing the severity of ARDS are therefore the number 1 target for COVID-19 therapy.

Neutrophils in ARDS Neutrophil influx into the extravascular compartments of the lungs is a defining characteristic of ARDS. During ARDS, circulating neutrophils become primed, resulting in reduce deformability and retention within the pulmonary capillary bed. They then migrate across the endothelium through the interstitium and epithelium into the airways themselves. As neutrophils migrate they are activated and release oxidants, proteases and neutrophil extracellular traps. All of these processes are important in killing bacterial pathogens but in ARDS these processes become prolonged and excessive leading to progressive lung damage. Neutrophil elastase and other neutrophil proteases such as proteinase-3 and cathepsin-G cause tissue injury resulting in increased epithelial and endothelial permeability which leads to the influx of protein-rich alveolar oedema.

Mortality in ARDS correlates directly with the extent of neutrophilia in the lung. Both human clinical data and murine studies demonstrate a key role for neutrophils in ARDS. Neutrophil depletion in multiple models of ARDS including those induced by lipopolysaccharide, acid, ventilator lung injury, transfusion and other stimuli, reduces the severity of acute lung injury including endothelial-epithelial cell damage and capillary-alveolar permeability.

Neutrophil proteases and particularly neutrophil elastase are believed to be central to the neutrophil induced lung damage. Neutrophil elastase is a serine protease contained within primary neutrophil granules which is released in response to neutrophil activation or neutrophil extracellular trap formation. It is involved in the pathogenesis of multiple inflammatory diseases and therapeutic development of neutrophil elastase inhibitors for use in ARDS has been ongoing for many years. Neutrophil elastase is markedly elevated in human ARDS samples and the inhibition of neutrophil elastase has been demonstrated to reduce epithelial injury in multiple animal models of lung injury across multiple stimuli including lipopolysaccharide (LPS), bleomycin, ventilation, sepsis and many others. Neutrophil elastase is critical to the development of neutrophil extracellular traps, which are highly damaging webs of DNA studded with proteases and other neutrophil derived toxins. Neutrophil extracellular traps (NET) formation and the failure to clear NETs have been strongly implicated in the development and poor outcomes from ARDS. Inhibition of neutrophil elastase reduces the formation of NETs.

A challenge therapeutically has been how to inhibit neutrophil elastase since administration of competitive inhibitors either orally or through the inhaled route may not be sufficient to block elastase activity in the lung.

RATIONALE Neutrophil elastase, proteinase-3 and cathepsin-G are activated during neutrophil maturation in the bone marrow through dipeptidyl peptidase 1 (DPP1; also known as cathepsin C), which removes the N-terminal dipeptide sequence of neutrophil serine proteases allowing active enzymes to be packaged into granules prior to release of neutrophils into the circulation. Brensocatib (INS1007, formerly AZD7986) is an orally delivered selective, competitive, and reversible inhibitor of DPP1. Brensocatib has been shown to inhibit neutrophil serine protease activity in blood in both animal models and healthy volunteers.

The investigators recently conducted a large phase 2 study of Brensocatib in patients with bronchiectasis designed to test if treatment with Brensocatib could reduce infective exacerbations and reduce neutrophil elastase activity in the lung in bronchiectasis patients. The study met its primary endpoint of time to first exacerbation and key secondary endpoint of the frequency of exacerbations as well as showing marked reductions in neutrophil elastase concentrations in sputum. Due to the need to replace the circulating pool of neutrophils with new neutrophils which are deficient in elastase, Brensocatib does not have its effect immediately, but rather over several days. Elastase concentrations were reduced at the first time point at day 14 in the phase 2 study, with very large reductions observed at the second time point at day 28.

In a cohort of 191 hospitalised COVID-19 patients with a completed outcome, the median time from illness onset to discharge was 22·0 days (IQR 18·0-25·0) and the median time to death was 18·5 days (15·0-22·0). Thirty-two patients (17%) required invasive mechanical ventilation and the median time from onset to mechanical ventilation was 14.5 days. The investigators hypothesise that the mechanism of action of Brensocatib to reduce protease activity will be more rapid in COVID-19 patients compared to bronchiectasis due to a more rapid turnover of neutrophils in acute illness. The objective is to test whether by reducing neutrophil protease activity in neutrophils the investigatorscan prevent or reverse the development of ARDS and thereby improve outcomes in individuals with COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

6.1. Inclusion criteria

• Male or female

* ≥16 years of age
* SARS-CoV-2 infection (clinically suspected+ or laboratory confirmed*).
* Admitted to hospital as in-patient less than 96 hours prior to randomisation^
* Illness of any duration, and at least one of the following:

  * Radiographic infiltrates by imaging (e.g. chest x-ray, computed tomography (CT) scan) OR
  * Evidence of rales/crackles on physical examination OR
  * Peripheral capillary oxygen saturation (SpO2) ≤94% on room air prior to randomization OR
  * Requiring supplemental oxygen. OR
  * Lymphocyte count <1 x 109 cells per litre (L)
* Participant (or legally authorized representative) provides written informed consent
* Able to take oral medication
* Participant (or legally authorised representative) understands and agrees to comply with planned trial procedures.

  * Laboratory-confirmed: SARS-CoV-2 infection as determined by polymerase chain reaction (PCR), or other commercial or public health assay in any specimen < 96 hours prior to randomization.

    * Clinically suspected: in general, SARS-CoV-2 infection should be suspected when a patient presents with (i) typical symptoms (e.g. influenza-like illness with fever and muscle pain, or respiratory illness with cough and shortness of breath); and (ii) compatible chest X-ray findings (consolidation or ground-glass shadowing); and (iii) alternative causes have been considered unlikely or excluded (e.g. heart failure, influenza). However, the diagnosis remains a clinical one based on the opinion of the managing doctor

      * Where a patient has been admitted to hospital for a non COVID-19 reason and develops COVID-19 symptoms whilst an in-patient, randomisation may occur up to 96 hours from onset of symptoms.

Exclusion Criteria:

* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 5 times the upper limit of normal, result within 72 hours of randomization (the result closest to randomization should be used if several results are available).
* History of severe liver disease
* Stage 4 severe chronic kidney disease or requiring dialysis (i.e. estimated Glomerular Filtration Rate < 30), result within 72 hours of randomization (the result closest to randomization should be used if several results are available)
* Absolute neutrophil count less than 1.0 x 109 cells per L within 72 hours of randomization (the result closest to randomization should be used if several results are available)
* Current treatments with potent Cyp3A4 inducers/inhibitors (e.g Itraconazole, Ketoconazole, diltiazem, verapamil, phenytoin or rifampicin)
* HIV treatments - current treatment with protease/integrase inhibitors or non-nucleoside reverse transcriptase inhibitors*
* Pregnant or breast feeding.
* Anticipated transfer to another hospital which is not a trial site within 24 hours.
* Allergy to Brensocatib
* Use of any investigational drug within five times of the elimination half-life after the last trial dose or within 30 days, whichever is longer. Co-enrolment with COVID-19 trials is allowed as per co-enrolment agreements and/or individual decision by the Chief Investigator.

Women of child-bearing potential must be willing to have pregnancy testing prior to trial entry.

*The Liverpool HIV checker (https://www.hiv-druginteractions.org/checker) should be used to check for any HIV drug interactions. Simvastatin could be used as a surrogate for Brensocatib as it metabolised similarly by CYP 3A4 pathway.

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 406 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Chalmers, Principal Investigator — University of Dundee
Locations (16):
- United Kingdom (16):
  - NHS Grampian, Aberdeen
  - Royal United Hospitals Bath NHS Foundation Trust, Bath
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Cardiff & Vale University Health Board, Cardiff
  - NHS Tayside, Dundee
  - NHS Fife, Dunfermline
  - Frimley Health NHS Foundation Trust, Frimley
  - Princess Alexandra Hospital NHS Trust, Harlow
  - NHS Highland, Inverness
  - NHS Forth Valley, Larbert
  - University Hospitals of Leicester NHS Trust, Leicester
  - Liverpool University Hospitals NHS Foundation Trust, Liverpool
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Hospitals North Midlands NHS Trust, Stoke-on-Trent
  - NHS Lanarkshire, Wishaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This double-blind, randomized, parallel-group, placebo-controlled trial was conducted at 14 secondary care sites in the United Kingdom Between 05th June 2020 and 28 February 2021
Pre-assignment Details: There were two post-randomisation exclusions due to ineligibility in the Brensocatib arm (one was admitted to hospital as an in-patient more than 96 hours prior to randomisation and another was receiving a prohibited medication). These two patients were included in the safety analysis. Four hundred and four participants (190 Brensocatib and 214 placebo) were included in the intention-to-treat analysis.
Groups:
- Brensocatib: Brensocatib oral tablet, 25mg once per day for 28 days
  Brensocatib: Selective, competitive, and reversible inhibitor of Dipeptidyl peptidase-1 (DPP1)
Period: Overall Study
Arm/Group | Brensocatib | Placebo
Started | 192 | 214
Completed | 187 (Participants with data for the primary outcome) | 211 (Participants with data for the primary outcome)
Not Completed | 5 | 3
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intention to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | Brensocatib | Placebo | Total
Number analyzed (Participants) | 190 | 214 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (12.5) | 62.0 (14.9) | 62.2 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 87 | 152
  Male | 125 | 127 | 252
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 11 | 20
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 175 | 195 | 370
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 5 | 4 | 9
Chronic cardiac disease [Count of Participants; unit: Participants] | 34 | 37 | 71
COPD [Count of Participants; unit: Participants] | 29 | 22 | 51
Obesity [Count of Participants; unit: Participants] | 41 | 48 | 89
Diabetes without complications [Count of Participants; unit: Participants] | 29 | 33 | 62
Hospitalized, not requiring supplemental oxygen [Count of Participants; unit: Participants] | 42 | 50 | 92
Hospitalized, requiring supplemental oxygen [Count of Participants; unit: Participants] | 128 | 140 | 268
Hospitalized, on non-invasive ventilation or high flow oxygen devices [Count of Participants; unit: Participants] | 20 | 24 | 44

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Participant Clinical Status Between Treatment Arms
Description: To determine the participant clinical status on a 7-point ordinal scale, minimum value 1, maximum value 7. Higher values indicate a worse outcome:
  1. Not hospitalised, no limitations on activities
  2. Not hospitalised, limitation on activities;
  3. Hospitalised, not requiring supplemental oxygen;
  4. Hospitalised, requiring supplemental oxygen;
  5. Hospitalised, on non-invasive ventilation or high flow oxygen devices;
  6. Hospitalised, on invasive mechanical ventilation or Extracorporeal membrane oxygenation (ECMO)
  7. Death.
Time Frame: Up to 29 days
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 187 | 211
participants
  Not hospitalized, no limitations on activities | 28 | 40
  Not hospitalized, limitations on activities | 112 | 129
  Hospitalized, not requiring supplemental oxygen | 7 | 11
  Hospitalized, requiring supplemental oxygen | 6 | 1
  Hospitalized, on non-invasive ventilation or high flow oxygen devices | 0 | 1
  Hospitalized, on invasive mechanical ventilation or ECMO | 5 | 6
  Death | 29 | 23
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; p = 0.008, Odds ratio Ordinal Logistic Regression; adjusted for the stratifying factors of age as a fixed effect and site using robust standard errors to account for clustering; Odds Ratio (OR) = 0.72, 95% CI 2-sided [0.57 to 0.92]

2. Secondary Outcome: Improvement of One Category From Admission Using 7-point Ordinal Scale.
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: 7-point ordinal scale, minimum value 1, maximum value 7. Higher values indicate a worse outcome:
  1. Not hospitalised, no limitations on activities
  2. Not hospitalised, limitations on activities
  3. Hospitalised, not requiring supplemental oxygen
  4. Hospitalised, requiring supplemental oxygen
  5. Hospitalised, on non-invasive ventilation or high flow oxygen devices
  6. Hospitalised, on invasive mechanical ventilation or Extracorporeal membrane oxygenation (ECMO)
  7. Death
Time Frame: Day 29
Population: ITT. Days to improvement was derived as
  1. days from randomization to date of first follow-up day where there was an improvement in CSTAT
  2. those who died before improvement were censored at date of death.
  3. those who withdrew or were loss to follow-up before improvement, if their day 29 status was unknown, they were censored at the date of loss to follow-up/withdrawal
  4. other participants were censored at day 29 from randomisation in study time if there were no improvement.
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
Participants | 159 | 186
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; p = 0.058, Regression, Cox; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.76 to 1.00]

3. Secondary Outcome: Participant Clinical Status on 7-point Ordinal Scale
Description: as for outcome 2
Time Frame: Day 15
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
Participants
  Not hospitalised, no limitations on activities | 22 | 26
  Not hospitalised, limitations on activities | 103 | 124
  Hospitalised, not requiring supplemental oxygen | 12 | 19
  Hospitalised, requiring supplemental oxygen | 16 | 13
  Hospitalised, on non-invasive ventilation or high flow oxygen devices | 3 | 5
  Hospitalised, on invasive mechanical ventilation or ECMO | 9 | 6
  Death | 20 | 18
  Missing | 5 | 3

4. Secondary Outcome: Mean Change in the 7-point Ordinal Scale
Description: as for outcome 2
Time Frame: Baseline to days 3, 5, 8, 11 and 29
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on WHO scale
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
Units on WHO scale
  Baseline to day 29 | 1.0 (2.0) | 1.3 (2.0)
  Baseline to day 15 | 1.0 (1.8) | 1.2 (1.6)
  Baseline to day 11 | 0.9 (1.6) | 1.1 (1.5)
  Baseline to day 8 | 0.7 (1.5) | 0.9 (1.0)
  Baseline to day 5 | 0.5 (1.1) | 0.5 (1.1)
  Baseline to day 3 | 0.2 (0.8) | 0.2 (0.9)

5. Secondary Outcome: Number of Participants Discharged or to a National Early Warning Score (NEWS) of Equal or Less Than 2 and Maintained for 24 Hours, Whichever Occurs First.
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: National Early Warning Score (NEWS). NEWS is a system that scores 6 physiological parameters (respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness or new-onset confusion, temperature) to give an aggerate score. Minimum score is 1, maximum score is 20.. Higher scores indicate worsening clinical outcomes.
Time Frame: Up to 29 days
Population: ITT. Those who died before being discharged or having a NEWS of ≤ 2 were censored at date of death. For those who withdrew or were loss to follow-up before being discharged or having a NEWS of ≤ 2, if their day 29 status was unknown, they were censored at the date of loss to follow-up/withdrawal. Other participants were censored at day 29 or 28 days from randomisation in study time if they were still in hospital and never had a NEWS of ≤ 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
Participants | 172 | 195
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.84 to 1.13]

6. Secondary Outcome: Change From Baseline of National Early Warning Score (NEWS).
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: National Early Warning Score. NEWS is a system that scores 6 physiological parameters (respiration rate, oxygen saturation, systolic blood pressure, pulse rate, level of consciousness or new-onset confusion, temperature) to give an aggerate score. Minimum score is 1, maximum score is 20.. Higher scores indicate worsening clinical outcomes.
Time Frame: Baseline to day 15
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
Participants
  -11 | 1 | 0
  -9 | 2 | 0
  -8 | 0 | 1
  -7 | 1 | 0
  -6 | 0 | 2
  -5 | 1 | 0
  -4 | 1 | 3
  -3 | 4 | 1
  -2 | 1 | 1
  -1 | 3 | 3
  0 | 15 | 24
  1 | 22 | 24
  2 | 36 | 34
  3 | 28 | 36
  4 | 21 | 28
  5 | 10 | 14
  6 | 11 | 6
  7 | 3 | 4
  8 | 1 | 4
  9 | 0 | 2
  10 | 0 | 1
  missing | 29 | 26

7. Secondary Outcome: Number of Oxygen Therapy Free Days
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: oxygenation
Time Frame: 1-29 days
Population: ITT.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
days | 24 [11 to 27] | 24.5 [17 to 27]
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Rate ratio = 0.93, 95% CI 2-sided [0.87 to 0.99]

8. Secondary Outcome: Incidence and Duration of New Oxygen Therapy Use During the Trial
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: oxygenation
Time Frame: 0-29 days
Population: For the duration of new oxygen use analysis, only participants who were hospitalised but not requiring supplemental oxygen (CSTAT = 3) at baseline were included
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 39 | 42
days | 0 [0 to 2] | 0 [0 to 1]
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Rate ratio = 1.13, 95% CI 2-sided [0.73 to 1.74]

9. Secondary Outcome: Number of Mechanical Ventilator Free Days
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: Mechanical ventilation
Time Frame: 1-29 days
Population: ITT
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
days | 28 [22 to 28] | 28 [26 to 28]
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Rate ratio = 0.84, 95% CI 2-sided [0.69 to 1.04]

10. Secondary Outcome: Incidence and Duration of New Mechanical Ventilation Use During the Trial.
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: Mechanical ventilation
Time Frame: 1-29 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
days | 0 [0 to 0] | 0 [0 to 0]
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Rate ratio = 1.68, 95% CI 2-sided [1.09 to 2.58]

11. Secondary Outcome: Duration of Hospitalisation (Days).
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: hospitalisation
Time Frame: Duration between date of admission and discharge assessed up to 29 days.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
days | 8.4 (8.3) | 8.2 (8.3)
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Rate ratio = 1.03, 95% CI 2-sided [0.92 to 1.15]

12. Secondary Outcome: 28-day Mortality
Description: Evaluation of the clinical efficacy of Brensocatib relative to standard care: mortality. Survival analysis was used to compare 28-day mortality between the treatment arms. Participants who did not die were censored on the last study day. Those who withdrew or were loss to follow-up and their day 29 status was unknown were censored at the date of loss to follow-up/withdrawal. Other participants were censored 28 days from randomisation in study time.
Time Frame: Day 1 to 29
Population: ITT
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
Participants | 29 | 23
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.41, 95% CI 2-sided [1.06 to 1.88]

13. Secondary Outcome: Cumulative Incidence of Serious Adverse Events (SAEs)
Description: Evaluation of the safety of the intervention through 29 days of follow-up as compared to the control arm
Time Frame: 1-29 days
Population: There were two post-randomisation exclusions due to ineligibility in the brensocatib group (one patient was admitted to hospital as an inpatient more than 96 h before randomisation and another was receiving a prohibited medication). These 2 excluded patients were included with the ITT population in the safety analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 192 | 214
Participants | 40 | 35

14. Secondary Outcome: Discontinuation or Temporary Suspension of Treatment
Description: Evaluation of the safety of the intervention through 28 days of follow-up as compared to the control arm
Time Frame: 1-29 days
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 192 | 214
Participants | 13 | 12

15. Secondary Outcome: Changes in White Cell Count (x10^9/L) Over Time (Hospitalised Participants Only)
Description: Evaluation of the safety of the intervention through 28 days of follow-up as compared to the control arm
Time Frame: Day 29
Population: Hospitalised participants only
Measure: Mean (Standard Deviation); unit: 10^9cells/L
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 14 | 18
10^9cells/L | 8.9 (4.7) | 8.5 (3.1)

16. Secondary Outcome: Changes in Haemoglobin (g/L) Over Time (Hospitalised Participants Only)
Description: Evaluation of the safety of the intervention through 28 days of follow-up as compared to the control arm
Time Frame: Day 29
Population: Hospitalised participants only
Measure: Mean (Standard Deviation); unit: g/l
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 14 | 18
g/l | 195.4 (264) | 105.5 (21.7)

17. Secondary Outcome: Changes in Platelets (x10^9/L) Over Time (Hospitalised Participants Only)
Description: Evaluation of the safety of the intervention through 28 days of follow-up as compared to the control arm
Time Frame: Day 29
Population: Safety
Measure: Mean (Standard Deviation); unit: 10^9cells/L
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 14 | 18
10^9cells/L | 270 (94.3) | 269 (117)

18. Secondary Outcome: Changes in Creatinine (Umol/L) Over Time (Hospitalised Participants Only)
Description: Evaluation of the safety of the intervention through 28 days of follow-up as compared to the control arm
Time Frame: Day 29
Population: Hospitalised patients only
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 14 | 19
umol/L | 84.9 (39) | 84.1 (52)

19. Secondary Outcome: Changes in Total Bilirubin (Umol/L) Over Time (Hospitalised Participants Only)
Description: Evaluation of the safety of the intervention through 28 days of follow-up as compared to the control arm
Time Frame: Day 29
Population: Safety
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 14 | 16
umol/L | 8.4 (3.9) | 9.3 (9.8)

20. Secondary Outcome: Changes in Alanine Aminotransferase (U/L) Over Time (Hospitalised Participants Only)
Description: Evaluation of the safety of the intervention through 28 days of follow-up as compared to the control arm
Time Frame: Day 29
Population: safety
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 14 | 15
U/L | 62.8 (43.2) | 52.3 (92.8)

21. Secondary Outcome: Changes in Aspartate Aminotransferase U/L Over Time (Hospitalised Participants Only)
Description: Evaluation of the safety of the intervention through 28 days of follow-up as compared to the control arm
Time Frame: Day 29
Population: Safety
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 3 | 4
U/L | 22 (11.4) | 28.8 (14.9)

22. Secondary Outcome: Adverse Events of Special Interest- Hyperkeratosis, Infections and Dental Complications
Description: Evaluation of the safety of the intervention through 29 days of follow-up as compared to the control arm
Time Frame: 1-29 days
Population: Safety
Measure: Count of Participants; unit: Participants
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 192 | 214
Participants
  Hyperkeratosis | 0 | 0
  Dental complications | 0 | 1
  Secondary infections | 6 | 7

23. Other Pre Specified Outcome: Percent of Participants With SARS-CoV-2 Detectable in Nasopharyngeal Sample
Description: Evaluation of the virologic efficacy of Brensocatib by assessing percent of participants with SARS-CoV-2 detectable in nasopharyngeal sample
Time Frame: Day 15 and day 29
Reporting Status: Not Posted

24. Other Pre Specified Outcome: Quantitative SARS-CoV-2 Virus in Nasopharyngeal Samples.
Description: Evaluation of the virologic efficacy of Brensocatib by assessing presence of SARS-CoV-2 virus in nasopharyngeal samples
Time Frame: Day 15 and day 29
Reporting Status: Not Posted

25. Other Pre Specified Outcome: Neutrophil Elastase and Heparin Binding Protein Measurement in Blood
Description: Evaluation of the virologic efficacy of Brensocatib by measuring neutrophil elastase and heparin binding protein measurement in blood
Time Frame: Days 1, 8, 15, 29
Reporting Status: Not Posted

26. Other Pre Specified Outcome: Blood Neutrophil Elastase Activity
Description: Neutrophil elastase activity was measure as follows: whole blood samples were treated with either 10mg/mL zymosan to stimulate neutrophil degranulation or with hanks' balanced salt solution (HBSS) at 37°C for 30 minutes. Following incubation, samples were centrifuged, and blood plasma frozen at -80°C for analysis. Neutrophil elastase activity was subsequently measured by cleavage of the specific fluorogenic substrate MeOSuc-AAPV-AMC. The stimulated elastase activity was calculated by subtracting the plasma elastase activity following incubation with zymosan stimulation from the elastase activity after incubation with buffer alone. Results presents arbitrary fluorescence intensity units (units/mL) as no reference standard is included in the assay. This outcome was included to assess the inhibition of neutrophil serine proteases by DPP1 treatment. Lower values indicate reduced elastase activity.
Time Frame: Day 29
Population: Substudy
Measure: Mean (Standard Deviation); unit: Units/ml
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 50 | 48
Units/ml | 103 (65) | 166 (97)
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Mean Difference (Final Values) = -67, 95% CI 2-sided [-102 to -31]

27. Other Pre Specified Outcome: Neutrophil Extracellular Trap Release
Description: Evaluation of the virologic efficacy of Brensocatib
Time Frame: Days 1, 15, 29
Reporting Status: Not Posted

28. Other Pre Specified Outcome: Neutrophil Surface Protein Expression Analysis
Description: Evaluation of the virologic efficacy of Brensocatib by flow cytometry- CD88, CXCR2, CD66b, CD11b, CD63)
Time Frame: Days 1, 15, 29
Reporting Status: Not Posted

29. Other Pre Specified Outcome: Neutrophil Phagocytosis of FITC-labelled Bacteria by Flow Cytometry
Description: Evaluation of the virologic efficacy of Brensocatib by flow cytometry
Time Frame: Days 1, 15, 29
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Quality of Life Measured by EuroQol-5 Dimensions-5 Levels (EQ-5D-5L)
Description: To evaluate patient reported outcome measures between the groups using EQ-5D-5L questionnaire. EQ-5D-5L comprises of five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and each dimension has 5 levels. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state. The total EQ-5D-5L score ranges from -0.594 to 1. A higher total score indicates better outcome.
Time Frame: Day 29
Population: ITT
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brensocatib | Placebo
Number analyzed (Participants) | 190 | 214
units on a scale | 0.67 (0.29) | 0.67 (0.25)
Statistical Analysis 1: Comparison: Brensocatib vs Placebo; Test type: Superiority; Mean Difference (Final Values) = 0.003, 95% CI 2-sided [-0.06 to 0.066]

ADVERSE EVENTS:
Time Frame: 29 days
Description: Adverse events were reported by the participant, site principal investigators or delegated staff responsible for detecting documenting and recording events that met the definition of an adverse event. Participants discharged from hospital before the end of the trial were given a diary to record adverse events up to day 28. Site principal investigators were responsible for assigning seriousness and causality of AEs
Arm/Group | Brensocatib | Placebo
All-Cause Mortality (participants affected / at risk) | 29/192 | 23/214
Serious Adverse Events (participants affected / at risk) | 40/192 | 35/214
Other Adverse Events (participants affected / at risk) | 86/192 | 99/214
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brensocatib (N=192) | Placebo (N=214)
Cardiac disorders (Cardiac disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders (Gastrointestinal disorders) | 1 (1) | 3 (3)
General disorders (General disorders) | 1 (1) | 0 (0)
Infections (Infections and infestations) | 26 (26) | 23 (23) — Including COVID-19
Neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Nervous system disorders (Nervous system disorders) | 4 (4) | 2 (2)
Psychiatric disorders (Psychiatric disorders) | 0 (0) | 2 (2)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 5 (5)
Skin disorders (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Vascular disorders (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brensocatib (N=192) | Placebo (N=214)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 4 (4)
Cold sweat (General disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 2 (2) | 0 (0)
Swelling face (General disorders) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Hallucination, visual (Psychiatric disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Nightmare (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (2) | 2 (4)
Liver function test abnormal (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Blood glucose abnormal (Investigations) | 1 (1) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Tachyarrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 5 (5)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral mucosal eruption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glossodynia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Tongue blistering (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oral mucosal blistering (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen tongue (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hypoaesthesia oral (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue erythema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) — Pruritis soles of feet
Rash pustular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 5 (5) | 7 (7)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Mouth ulceration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Widespread surgical emphysema in arms and neck, shown in CXR.
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2)
Oral candidiasis (Infections and infestations) | 0 (0) | 3 (3)
Candida infection (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Vulvovaginal candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Serratia infection (Infections and infestations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Steroid diabetes (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Undiagnosed Diabetes (new presentation) - steroid induced
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/32/NCT04817332/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-05): https://cdn.clinicaltrials.gov/large-docs/32/NCT04817332/SAP_001.pdf